CLINICAL TRIAL: NCT03022279
Title: Transversus Abdominis Plane Block vs. Local Wound Infiltration for Elective Laparoscopic Cholecystectomy in Children and Adolescents: A Prospective Randomized-Controlled Trial
Brief Title: Nerve Blocks vs Local Injections for Post-op Pain Prevention in Laparoscopic Cholecystectomy in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brian Wallace Gray (Other)
Responsible Party: Sponsor-Investigator, Brian Wallace Gray, Pediatric surgeon, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1410511719
Record Dates: First submitted 2016-11-25; First posted 2017-01-16 (Estimated); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Pediatric; post-operative pain prevention; Anesthesia, Infiltration; Nerve Blockade
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP blocks (Active Comparator): TAP block group will receive three injections performed by an Anesthesiologist trained in the procedure, prior to initiation of the surgical procedure. Bilateral posterior transversalis fascial plane blocks and a right sided subcostal transverse abdominal plane block will be placed under ultrasound guidance. Normal saline will be used to confirm proper muscle layer placement before instillation of the local anesthesia. All patients will receive 2.5 mg/kg or 1 mL/kg of 0.2% ropivacaine with maximum of 60 mL (divided equally amongst the injection sites).
  Interventions: Procedure: TAP Blocks
- Local Wound Infiltration (Active Comparator): Local wound infiltration (LWI) will be performed by the operative surgeon using 2.5 mg/kg or 1 mL/kg of 0.2% ropivacaine with maximum of 60 mL divided amongst the four port sites. 40% of the total dose will be given at the umbilicus, and 20% will be given at each of the other 3 ports. The majority of the anesthetic will be administered at the peritoneal level. Laparoscopic/robotic cholecystectomy will be performed with a port at the umbilicus and three smaller ports in a standard fashion in the subxiphoid and right upper quadrant regions. If conversion to open cholecystectomy occurs, the study data will still be collected, but the patient's data will be excluded from analysis.
  Interventions: Procedure: local wound infiltration

INTERVENTIONS:
Procedure: TAP Blocks — ultrasound guided transversus abdominis plane block utilizing 2.5 mg/kg or 1 mL/kg of 0.2% ropivacaine
  Other Names: nerve block; transversus abdominis plane block
  Arms: TAP blocks
Procedure: local wound infiltration — local anesthesia provided at the surgical site utilizing 2.5 mg/kg or 1 mL/kg of 0.2% ropivacaine
  Other Names: local wound injections
  Arms: Local Wound Infiltration

SUMMARY:
The objective of this study is to compare transversus abdominis plane (TAP) blocks to local wound infiltration (LWI) in terms of postoperative pain control in pediatric patients undergoing elective laparoscopic cholecystectomy. Our hypothesis is that TAP blocks will be superior to LWI for postoperative pain control resulting in decreased use of opioid / narcotic pain medication and decreased pain scored in the immediate 24-hour postoperative period. The rationale is that determining the effect of analgesia in this pediatric population is important to optimize clinical care.

DETAILED DESCRIPTION:
In this study, patients ages 8 through 17 years scheduled for elective laparoscopic cholecystectomy will be invited to participate. Those having da Vinci cholecystectomy procedures will also be eligible. The da Vinci System is a minimally invasive option utilizing robotic technology. Once randomized, the patient will undergo either ultrasound guided bilateral TAP blocks or LWI at the beginning of the surgical procedure. Prospective data regarding pain scores, use of opioid medication, and nausea and vomiting episodes will be collected for both groups. Due to the nature of the study, it will not be possible to blind the investigators to the randomly selected method of injecting local anesthesia; however the personnel involved in the post-anesthetic and post-operative assessment will be blinded to the intervention, as well as the subjects themselves.

ELIGIBILITY:
Inclusion Criteria:

1. 8-17 yrs of age at date of enrollment.
2. Elective laparoscopic or da Vinci cholecystectomy scheduled for any diagnostic reason.

Exclusion Criteria:

1. Chronic pain or chronic use of narcotic or other prescription pain medications.
2. Use of pain medication within 24 hours before surgery
3. Prior major abdominal surgery
4. Evidence of acute inflammation
5. Patients with acute cholecystitis
6. Bleeding / coagulation disorder
7. Seizure disorder
8. Renal dysfunction
9. Infection at injection sites for TAP block or trocar placement
10. Contraindication to LWI or TAP block procedure, as determined by surgeon or anesthesiologist performing the procedure (including, but not limited to, previous incision distorting anatomy or inability to visualize anatomical planes)
11. Any known allergy to medications used in this study
12. Patient unable to verbalize pain score or independently assess pain level
13. Unstable patient in need of emergent intervention at surgeon discretion
14. Patients who are known to be pregnant
15. Patients who are currently prisoners
16. Children in custody of the state
17. Subjects will a BMI >/= 50
18. Investigator discretion for any other reason

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2022-09 (Actual); Study Completion 2022-09 (Actual)

PRIMARY OUTCOMES:
Amount of narcotic pain medication | 24 hours post-op
Time to first request of pain medication | From post-anesthesia care unit "(PACU) in" time to first pain medication dose, up to 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gray Brian, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children at IU Health, Indianapolis, Indiana, United States